CLINICAL TRIAL: NCT03214406
Title: Clinical Evaluation of the Efficacy of a Marketed Dentifrice on Plaque and Gingivitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Church & Dwight Company, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ST-7323
Record Dates: First submitted 2017-07-10; First posted 2017-07-11 (Actual); Results first posted 2019-07-23 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-04

CONDITIONS: Plaque; Gingivitis
MeSH Terms: conditions — Plaque, Amyloid; Gingivitis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Arm & Hammer Advance White Brilliant Sparkle (Test product) (Experimental): 2X daily brushing for 12 weeks with Arm & Hammer Advance White Brilliant Sparkle (Test product). Return to pre-study hygiene regimen for 4 weeks and final evaluation at 16 weeks.
  Interventions: Drug: Arm & Hammer Advance White Brilliant Sparkle (Test product)
- Crest Cavity Protection Regular Toothpaste (Negative Control) (Active Comparator): 2X daily brushing for 12 weeks with Crest Cavity Protection Regular Toothpaste (Negative Control). Return to pre-study hygiene regimen for 4 weeks and final evaluation at 16 weeks.
  Interventions: Drug: Crest Cavity Protection Regular Toothpaste (Negative Control)

INTERVENTIONS:
Drug: Arm & Hammer Advance White Brilliant Sparkle (Test product) — 20% sodium bicarbonate
  Arms: Arm & Hammer Advance White Brilliant Sparkle (Test product)
Drug: Crest Cavity Protection Regular Toothpaste (Negative Control) — Negative control
  Arms: Crest Cavity Protection Regular Toothpaste (Negative Control)

SUMMARY:
Parallel, double blind, randomized, Institutional Review Board (IRB) -approved study involving approximately 160 subjects to complete. Subjects were randomly assigned to either the test product (Arm & Hammer Advance White Brilliant Sparkle) or the control (Crest Cavity Protection Regular) based on baseline mean whole-mouth plaque and gingival scores and age.Subjects brushed with their assigned dentifrice two times (2X) daily and were evaluated for gingivitis, bleeding and plaque at Baseline and after 4-, 8-, and 12-weeks of product use. Return to pre-study hygiene regimen for 4 weeks and final evaluation at 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have provided written informed consent prior to being entered into study
* Have at least 18 scorable natural teeth as determined by the examiner
* Have a mean baseline plaque index score greater than or equal to 2.0 as determined by the Soparkar Modification of the Turesky modification of the Quigley-Hein Plaque Index
* Have a mean baseline gingival index score of greater than 1.80 as determined by the Modified Gingival Index
* Presence of greater than 10 bleeding sites upon probing
* Agree not to have dental prophylaxis or any other elective, no -emergency dental procedures (other than those provided during the study) any time during the study
* Agree to abstain from use of floss, chewing gum, mouth rinses, any toothpaste other than the study toothpaste, tooth whitening products (either professional or at home use) and all other oral hygiene other than the study procedures for the duration of the study.
* Agree to refrain from all oral hygiene on the morning of each evaluation visit and to refrain from eating and drinking for 4 hours prior to each evaluation visit
* Agree to comply with the conditions and schedule of the study

Exclusion Criteria:

* Physical limitations or restrictions that might preclude normal tooth brushing
* Evidence of gross oral pathology, including widespread caries or chronic neglect, extensive restoration, pre-existing gross plaque or soft or hard tissue tumor of the oral cavity.
* Heavy calculus that might interfere with evaluations as determined by the Investigator/Examiner
* Chronic disease with concomitant oral manifestations
* Conditions requiring antibiotic prophylaxis prior to invasive procedures, such as heart murmur, history of rheumatic fever, valvular disease or certain prosthetic implants
* History of uncontrolled diabetes or hepatic or renal disease, or other serious conditions or transmittable diseases (eg cardiovascular disease, AIDS)
* Subjects with fixed or removable orthodontic appliances or removable partial dentures
* Subjects who are currently undergoing, or require, extensive dental work or orthodontic treatment
* Treatment with antibiotics within the 1-month period before the baseline examination, or a condition that is likely to require antibiotic treatment over the course of the trial
* Chronic treatment (2 weeks or more) with any medication known to affect periodontal status (including phenytoin, calcium antagonists, cyclosporine, coumarin, nonsteroidal anti-inflammatory drugs, and aspirin) within 1 month of baseline examination. All other medications for chronic medical conditions must have been initiated at least 3 months before enrollment
* Moderately advanced to advanced periodontitis as indicated by clinical attachment loss, radiographic alveolar bone loss, and/or periodontal pockets greater than 5 millimeters
* Having history of early-onset periodontitis or acute necrotizing ulcerative gingivitis
* Concomitant endodontic or periodontal therapy other than prophylaxis in the last 6 months
* Professional prophylaxis within 1 month prior to the baseline clinical evaluation
* Currently using bleaching trays
* Currently using power toothbrush
* Currently a smoker or recently (during the past 6 months) quit smoking
* Having any oral piercings in or around the oral cavity with ornament or accessory
* Regular use of any chemotherapeutic antiplaque/antigingivitis products such as Colgate Total, Crest Pro-Health, Listerine, etc
* History of significant adverse effects following use of oral hygiene products such as toothpastes and mouthrinses
* Subjects who are nursing, pregnant or plan to become pregnant for the duration of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2010-02-08 (Actual); Primary Completion 2010-08-03 (Actual); Study Completion 2010-08-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- BioSci Research Canada, Ltd, Mississauga, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm & Hammer Advance White Brilliant Sparkle (Test Product): 2X daily brushing for 12 weeks with Arm & Hammer Advance White Brilliant Sparkle (Test product)
  Arm & Hammer Advance White Brilliant Sparkle (Test product): 20% sodium bicarbonate
- Crest Cavity Protection Regular Toothpaste (Negative Control): 2X daily brushing for 12 weeks with Crest Cavity Protection Regular Toothpaste (Negative Control)
  Crest Cavity Protection Regular Toothpaste (Negative Control): Negative control
Period: Overall Study
Arm/Group | Arm & Hammer Advance White Brilliant Sparkle (Test Product) | Crest Cavity Protection Regular Toothpaste (Negative Control)
Started | 88 | 93
Completed | 78 | 78
Not Completed | 10 | 15
Not completed — did not meet enrollment criteria | 9 | 13
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm & Hammer Advance White Brilliant Sparkle (Test Product) | Crest Cavity Protection Regular Toothpaste (Negative Control) | Total
Number analyzed (Participants) | 78 | 78 | 156
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 78 | 78 | 156
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 51 | 107
  Male | 22 | 27 | 49
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Gingvial Efficacy [Mean (Standard Deviation); unit: units on a scale] — Lobene Modified Loe-Silness Gingival Scoring Index (MGI) - gingival sites were visually scored at each visit on the buccal and lingual marginal gingivae and interdental papillae of all scorable teeth, using a scale of 0-4. Lower values represent a better outcome.
  units on a scale | 2.039 (.053) | 2.039 (.057) | 2.039 (.055)
Gingival Bleeding Efficacy [Mean (Standard Deviation); unit: units on a scale] — Bleeding was assessed on all scorable buccal and lingual surfaces by inserting a periodontal probe into the gingival crevice and sweeping from the distal aspect to the mesial aspect around the tooth at a depth of approximately 1 mm and angle of approximately 60 degrees while in contact with the sulcular epithelium. Three areas (distobuccal, midbuccal and midlingual) were assessed around each tooth. Sites were scored at each visit using the Gingival Bleeding Index (GBI) as defined by Saxton and van der Ouderaa on a scale of 0-2. Lower values represent a better outcome.
  units on a scale | .228 (.046) | .230 (.044) | .229 (.045)
Plaque Efficacy [Mean (Standard Deviation); unit: units on a scale] — Plaque was scored at each visit using the Soparker modification of the Turesky Modification of the Quigley-Hein Plaque Index (PI) on all scorable buccal and lingual surfaces. Plaque was stained with disclosant and each tooth was divided into six areas for scoring on a scale of 0-5. A PI score for each subject was calculated by adding all individual site scores (6 per tooth) and dividing by the total number of sites scored (teeth x 6). Lower values represent a better outcome.
  units on a scale | 2.575 (.295) | 2.534 (.248) | 2.555 (.272)

OUTCOME MEASURES:

1. Primary Outcome: Within-Treatment Whole-Mouth Differences (vs Baseline) - Gingival Efficacy
Description: change in score as measured by Gingival Index (0=absence of inflammation, 1=mild inflammation: slight change in color, little change in texture of any portion of but not the entire marginal or papillary gingival unit, 2=mild inflammation: slight change in color, little change in texture to entire marginal or papillary gingival unit, 3=moderate inflammation: glazing, redness, edema and/or hypertrophy of the marginal or papillary gingival unit, 4=severe inflammation: marked redness, edema and/or hypertrophy of the marginal or papillary gingival unit, spontaneous bleeding, congestion, or ulceration. The scale ranges from 0-4.
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm & Hammer Advance White Brilliant Sparkle (Test Product) | Crest Cavity Protection Regular Toothpaste (Negative Control)
Number analyzed (Participants) | 78 | 78
units on a scale
  4 weeks | .230 (.105) | .155 (.123)
  8 weeks | .3701 (.130) | .205 (.077)
  12 weeks | .444 (.139) | .214 (.110)
  16 weeks | .330 (.118) | .157 (.084)

2. Primary Outcome: Within-Treatment Whole-Mouth Differences (vs Baseline) Gingival Bleeding Efficacy
Description: change in score as measured by Gingival Bleeding Index (0=absence of bleeding after 30 seconds, 1= bleeding observed after 30 seconds, 2= bleeding occurs instantly). The scale ranges from 0-2.
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm & Hammer Advance White Brilliant Sparkle (Test Product) | Crest Cavity Protection Regular Toothpaste (Negative Control)
Number analyzed (Participants) | 78 | 78
units on a scale
  4 weeks | .134 (.055) | .119 (.056)
  8 weeks | .162 (.042) | .145 (.039)
  12 weeks | .190 (.045) | .162 (.056)
  16 weeks | .180 (.043) | .144 (.056)

3. Primary Outcome: Within-Treatment Whole-Mouth Differences (vs Baseline) - Plaque Efficacy
Description: change in score as measured by Plaque Index (0=no visible plaque, 1=separate flecks of plaque at the cervical margin of the tooth, 2=a thin, continuous band of plaque (up to 1mm wide) at the cervical margin, 3= a band of plaque wider than 1 mm but covering less than one-third of the crown, 4=plaque covering at least one-third but less than two-thirds of the crown, 5= plaque covering two-thirds or more of the crown. The scale ranges from 0-5.
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm & Hammer Advance White Brilliant Sparkle (Test Product) | Crest Cavity Protection Regular Toothpaste (Negative Control)
Number analyzed (Participants) | 78 | 78
units on a scale
  4 weeks | .648 (.327) | .468 (.264)
  8 weeks | .776 (.369) | .574 (.283)
  12 weeks | .765 (.295) | .533 (.332)
  16 weeks | .275 (.378) | .275 (.378)

ADVERSE EVENTS:
Arm/Group | Arm & Hammer Advance White Brilliant Sparkle (Test Product) | Crest Cavity Protection Regular Toothpaste (Negative Control)
Serious Adverse Events (participants affected / at risk) | 0/88 | 0/93
Other Adverse Events (participants affected / at risk) | 0/88 | 0/93

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Confidentiality agreement in place with Investigator.